CLINICAL TRIAL: NCT03175731
Title: A Randomized Controlled Study on the Effects of PPIs on Gastroesophageal Variceal Bleeding in Liver Cirrhosis (PPIs: Proton Pump Inhibitors)
Brief Title: PPIs and Gastroesophageal Varices in Liver Cirrhosis (PPIs: Proton Pump Inhibitors)
Acronym: PPIs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yanjing Gao (Other)
Responsible Party: Sponsor-Investigator, Yanjing Gao, Vice presidengt of Department of Gastroenterology of Qilu Hospital, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017037-QILU
Record Dates: First submitted 2017-05-25; First posted 2017-06-05 (Actual); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Liver Cirrhosis; Hypertension, Portal
Keywords: Gastroesophageal varices; Hemorrhage
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Hemorrhage | interventions — Proton Pump Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proton Pump Inhibitors (Experimental): Pantoprazole 40mg per day intravenously or orally for 2 weeks after endoscopic treatment.
  Interventions: Drug: Proton Pump Inhibitors
- Placebo (Placebo Comparator): Placebo 40mg per day intravenously or orally for 2 weeks after endoscopic treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proton Pump Inhibitors — Pantoprazole 40mg per day intravenously or orally for 2 weeks after endoscopic treatment.
  Other Names: Experimental
  Arms: Proton Pump Inhibitors
Drug: Placebo — Placebo 40mg per day intravenously or orally for 2 weeks after endoscopic treatment.
  Other Names: Control
  Arms: Placebo

SUMMARY:
This study is aimed at investigating the effect of PPIs on gastroesophageal varices in liver cirrhosis. Half of participants will receive PPI, while the other half will receive a placebo.

DETAILED DESCRIPTION:
PPIs can inhibit parietal cell H+/K+-ATPase and reduce secretion of gastric acid. PPIs can promote platelet aggregation and stabilize the formation of fibrin thrombosis by maintaining the high pH environment in the stomach and inactivating pepsin. The effect of PPIs on ulcerative upper gastrointestinal bleeding was confirmed but it is not clear whether PPIs is applicable in esophagogastric variceal bleeding whose etiology and bleeding position are different from ulcerative upper gastrointestinal bleeding. There is lack of consensus and sufficient evidences to support to use PPIs in esophagogastric variceal bleeding in cirrhotic patients universally. Nevertheless, the use of PPIs in liver cirrhotic patients with gastroesophageal varices is common.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cirrhosis
* GEVs was diagnosed by endoscopy

Exclusion Criteria:

* Acute gastrointestinal bleeding need emergency surgery
* Acid-related disease, such as peptic ulcer disease or gastroesophageal reflux diseases (GERD)
* Hepatocellular carcinoma (HCC) or other malignant tumor
* History of esophagus, stomach or liver surgery
* Child-Pugh C and can't be improved to Child-Pugh A or B
* Preparing to be pregnant, pregnant or breast feeding
* Allergic to PPIs(proton pump inhibitors) or intolerable
* Cannot provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing /A Gao, PhD.MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology,Qilu Hospital,Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Pump Inhibitors | Placebo
Started | 53 | 53
Completed | 46 | 48
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proton Pump Inhibitors | Placebo | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (10.0) | 54.2 (10.6) | 53.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 36 | 38 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Variceal Bleeding Events
Description: The primary endpoint was variceal bleeding, which was defined as hematemesis or melena from endoscopically proven GEVs, in the absence of any other lesion that might explain the bleeding.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Pump Inhibitors | Placebo
Number analyzed (Participants) | 53 | 53
Participants | 3 | 3

2. Secondary Outcome: Mortality
Description: Prognosis of esophagogastric variceal bleeding.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Pump Inhibitors | Placebo
Number analyzed (Participants) | 53 | 53
Participants | 1 | 0

3. Secondary Outcome: Adverse Eventsafter Endoscopic Therapy
Description: Advers events caused by endoscopic therapy, including chest pain, dysphagia, fever and so on
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Pump Inhibitors | Placebo
Number analyzed (Participants) | 53 | 53
Participants | 15 | 20

ADVERSE EVENTS:
Time Frame: 8 weeks after endoscopic therapy.
Arm/Group | Proton Pump Inhibitors | Placebo
All-Cause Mortality (participants affected / at risk) | 1/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 15/53 | 20/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Pump Inhibitors (N=53) | Placebo (N=53)
Chest discomfort (Gastrointestinal disorders) | 11 (11) | 14 (14)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT03175731/Prot_SAP_000.pdf